CLINICAL TRIAL: NCT05946044
Title: The Osteoarthritis Prevention Study
Acronym: TOPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Arthritis Foundation (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Disease Prevention (Unknown); Office of Research on Women's Health (ORWH) (NIH); Office of Behavioral and Social Sciences Research (OBSSR) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency); University of Missouri-Columbia (Other); Rapid Nutrition PLC (Unknown)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00080136; U01AR082121-01 (NIH)
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Obesity; Knee Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: assessor-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Control (No Intervention): This comparison group provides attention, social interaction, and healthy lifestyle classes. There will be 4, 1-hour face-to-face group meetings per year featuring community health professionals, quarterly newsletters, and quarterly text messages.
- Diet and Exercise (Experimental): The dietary component of the weight loss intervention is characterized by the frequency of contacts, methods to induce dietary restriction, and behavioral therapy strategies. The first 6 months of the diet program is an energy-restricted diet with the option of using partial meal replacements and nutritious snacks (Rapid Nutrition, PLC). The weight loss goal for the diet and exercise group is a minimum of 10% of baseline body weight by the end of year 1. The weight loss phase is followed by 3 years of a weight-loss maintenance program, with the goal of sustaining the achieved weight loss. The exercise component includes 60-minute sessions 2 days per week for 48 months.
  Interventions: Behavioral: Diet and Exercise

INTERVENTIONS:
Behavioral: Diet and Exercise — Group and individual weight loss and weight maintenance sessions combined with exercise throughout the 48 months.
  Arms: Diet and Exercise

SUMMARY:
The goal of this study is to establish the efficacy of an intervention of dietary weight loss, exercise, and weight-loss maintenance for knee Osteoarthritis (OA) prevention in adult females aged ≥ 50 years with obesity and no or infrequent knee pain. The primary aim is to compare the effects of a dietary weight loss, exercise, and weight-loss maintenance to an attention control group in preventing the development of structural Magnetic Resonance Imaging (MRI) knee OA. Secondary aims will determine the intervention effects on pain, mobility, health-related quality of life, knee joint compressive forces, inflammatory measures, weight loss, exercise self-efficacy, and cost-effectiveness of this intervention.

DETAILED DESCRIPTION:
Osteoarthritis (OA), the leading cause of disability among adults, is without a cure and is associated with significant comorbidities. OA ranks as the third most common diagnosis for hospital inpatient stays with 1.25 M per year, with the knee the most commonly affected weight-bearing joint. This study will address knee OA disease prevention in adult females because prevention of OA is preferable to treatment, females are affected at nearly twice the rate as males, and to date interventions designed to slow or stop knee OA progression have failed. Dietary weight loss, with and without exercise, has level 1 evidence of effective treatment for adults with knee OA and overweight and obesity. Reduced degenerative cartilage changes are also associated with weight loss, making it a possible preventive therapy for people at risk for knee OA. The objective of this Phase III, multi-site (Boston, MA, Chapel Hill, NC, Sydney, Australia, and Winston-Salem, NC) randomized clinical trial is to establish the efficacy of an intervention of dietary weight loss, exercise, and weight-loss maintenance for knee OA prevention. We will establish efficacy in structural, symptomatic, and mechanistic outcomes compared to attention control, and determine the cost-effectiveness of this non-pharmacologic, non-surgical intervention in preventing incident knee OA in adult females aged ≥ 50 years with obesity and no or infrequent knee pain, a cohort at high risk for knee OA.

Participants will be 1,230 ambulatory, community dwelling females with obesity (BMI ≥ 30 kg/m2), and aged ≥ 50 years. Structural and symptomatic eligibility will be determined at the individual knee level. The eligible knee will have no radiographic (Kellgren Lawrence (KL) score ≤ 1) and no MRI knee OA with no or infrequent knee pain (< 15 days/month) in the same knee. The primary aim is to compare the effects of a 48-month intervention of dietary weight loss, exercise, and weight-loss maintenance to an attention control group in preventing the development of structural (MRI) knee OA using the MRI OA Knee Score (MOAKS). Secondary aims will determine the intervention effects on the Knee Injury and Osteoarthritis Outcome Score (KOOS) pain, mobility (6 minute walk distance), and health-related quality of life (SF-36). Mechanistic secondary outcomes include knee joint compressive forces as a measure of joint loading, IL-6 as an inflammatory measure, and weight loss and exercise self-efficacy. A cost-effectiveness analysis will establish the value of the 48-month D+E (diet and exercise) intervention.

This study is significant in that it will test a critically needed primary prevention intervention of dietary weight loss, exercise, and weight-loss maintenance for females at risk for the development of knee OA designed to reduce incident structural knee OA compared to an attention control group, and intended to maximize health benefits at a reasonable cost.

ELIGIBILITY:
Inclusion Criteria:

* Female
* BMI ≥ 30 kg/m2
* An eligible knee will have no OA by xray and MRI
* No or infrequent knee pain (< 15 days/month) in the same knee

Exclusion Criteria:

* symptomatic or severe coronary artery disease
* unable to walk without a device
* blindness
* type 1 diabetes
* active treatment for cancer
* during the past 12 months knee fracture, anterior cruciate ligament (ACL), medial collateral ligament (MCL), or meniscus injury with or without surgical repair
* knee injection during the past 6 months
* bilateral knee OA by x-ray Kellgren-Lawrence (KL) ≥ 2
* bilateral knee OA by MRI
* bilateral symptomatic knee OA (frequent bilateral knee pain > 15 days per month)
* BMI< 30.0 kg/m2
* male sex
* claustrophobia
* contraindication to MRI including body weight > 300 lbs or knee coil does not fit
* unwillingness or inability to change eating and physical activity habits due to environment
* cannot speak and read English
* planning to leave area > 2 months during the 48-month intervention period

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1230 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Structural knee Osteoarthritis (OA) MRI change Scores | Month 48
  Compare the effects of a 48-month intervention of dietary weight loss, exercise, and weight-loss maintenance to an attention control group in preventing the development of structural (MRI) knee OA. Assessed using the MRI Osteoarthritis Knee Score (MOAKS). The MOAKS evaluates degenerative changes in the knee, including the location and severity of osteophyte formation, bone marrow lesions, and cartilage loss. The MOAKS classification system of osteophytes has grades ranging from 0 (none) to 3 (large).

SECONDARY OUTCOMES:
Knee Pain Scores | Month 48
  Compare the effects of a 48-month intervention of dietary weight loss, exercise and weight-loss maintenance to an attention control group on the Knee Injury and Osteoarthritis Outcome Score (KOOS pain). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score is calculated for the pain subscale. We will transform the score to a 0-100 scale, with 100 representing the most pain and 0 representing no pain.
Mobility Scores | Month 48
  Compare the effects of a 48-month intervention of dietary weight loss, exercise and weight-loss maintenance to an attention control group on 6-minute walk distance. Assessment of 6 minute walk distance (measured in meters). Greater distance indicates better mobility.
Health-Related Quality of Life Scores | Month 48
  Compare the effects of a 48-month intervention of dietary weight loss, exercise and weight-loss maintenance to an attention control group on health-related quality of life (SF-36). Questions from the SF-36 yield 2 broad summary scores: physical health and mental health. Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.

OTHER OUTCOMES:
Knee Joint Loading Number | Month 48
  Compare the effects of a 48-month intervention of dietary weight loss, exercise, and weight-loss maintenance to an attention control group on knee joint compressive loads (Newtons). Higher numbers indicate greater loads.
Inflammation Value | Month 48
  Compare the effects of a 48-month intervention of dietary weight loss, exercise, and weight-loss maintenance to an attention control group on plasma Interleukin-6 (IL-6). Higher values indicate more inflammation.
Self-Efficacy Scores - exercise | Month 48
  Compare the effects of a 48-month intervention of dietary weight loss, exercise, and weight-loss maintenance to an attention control group on exercise self-efficacy. Exercise self efficacy will be measured using the walking efficacy for duration scale measures one's ability to walk/jog at a moderately fast pace for various durations. Range 0-100. A higher score indicates a higher self-efficacy. indicate better self-efficacy.
Self-Efficacy Scores - weight loss | Month 48
  Compare the effects of a 48-month intervention of dietary weight loss, exercise, and weight-loss maintenance to an attention control group on weight loss self-efficacy. Weight-loss self efficacy will be measured by the weight efficacy lifestyle questionnaire. A 20-item measure developed to assess self-efficacy for weight management. Participants are asked to rate their confidence to resist the desire to eat using a 10-point scale ranging from 0 not confident to 9 very confident. Total scores range from 0-180. Higher scores indicate better self-efficacy.
Cost-Effectiveness Ratios | Month 48
  To establish the cost-effectiveness of this multimodal weight loss, exercise, and weight-loss maintenance program by conducting cost-effectiveness and budgetary impact analyses using data from the current trial in a validated computer-simulation model of knee OA. The cost-effectiveness ratio provides a measure of value for money. The cost-effectiveness of a specific prevention or treatment strategy is measured in dollars per quality-adjusted life-year gained ($/QALY). a budget impact analysis (BIA) of the weight loss program quantifies the financial consequences of adopting the weight loss program by various payer models.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Messier, Ph.D., Principal Investigator — Wake Forest University
Locations (4):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
- University of Sydney, Sydney, Australia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial after deidentification.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by the study P&P committee. Proposals should be directed to the study PI, Stephen Messier at messier@wfu.edu or the central contact.

REFERENCES:
- [Background] Messier SP, Callahan LF, Losina E, Mihalko SL, Guermazi A, Ip E, Miller GD, Katz JN, Loeser RF, Pietrosimone BG, Soto S, Cook JL, Newman JJ, DeVita P, Spindler KP, Runhaar J, Armitano-Lago C, Duong V, Selzer F, Hill R, Love M, Beavers DP, Saldana S, Stoker AM, Rice PE, Hunter DJ. The osteoarthritis prevention study (TOPS) - A randomized controlled trial of diet and exercise to prevent Knee Osteoarthritis: Design and rationale. Osteoarthr Cartil Open. 2023 Nov 20;6(1):100418. doi: 10.1016/j.ocarto.2023.100418. eCollection 2024 Mar. PMID 38144515